CLINICAL TRIAL: NCT02561637
Title: The SICAM-trial: Studying the Effect of Spouses' Involvement Through Case Management in Older Patients' Fast-track Program During and After Total Hip Replacement - A Quasi-experimental Study With a Complex Intervention
Brief Title: The Effect of Spouses' Involvement Through Case Management in Older Patients' Fast-track Program
Acronym: SICAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Connie Berthelsen, Assistant professor, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SICAM2015
Record Dates: First submitted 2015-09-21; First posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Case management
MeSH Terms: interventions — Case Management; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case management (Experimental): Before admission the spouse-patient dyads will take part in an interview with the case manager assessing the spouses' needs during admission through an individual care plan. During admission the case manager will follow-up and assess the goals and actions of the individual care plan and coordinate with other health professionals. During the discharge meeting the case manager will provide additional information to the spouse according to needs assessed in the care plan. After discharge the case manager will conduct a follow-up telephone call for the spouse 3-4 days and 10 days after the patient's discharge consisting of information similar to that provided at the discharge meeting.
  Interventions: Behavioral: Case management
- Control group (Other): Spouses and patients in the control group will receive usual care and written and oral information about the fast-track program and principles in general from the nursing staff. The usual care and information is provided before admission in the out-patient facilities and during admission
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Case management
  Arms: Case management
Behavioral: Control group
  Arms: Control group

SUMMARY:
Patients in fast-track programmes are required to take an active part in their treatment and rehabilitation. Spouses of older patients can often provide valued practical and emotional support, reducing stress, pain and length of stay - yet they are seldom invited to participate in a supporting role. The aim of this study is to investigate the effect of spouses' involvement in older patients fast-track treatment programs using case management as intervention. A two-group quasi-experimental design with pre-test and repeated post-test measures (protocol approved in November 2012) was used. Patients aged 65 years or older going through a fast-track programme for a total hip replacement and their spouses was recruited in dyads from one Danish orthopaedic ward for the intervention group (n=15) and for the control group (n=14). Data was collected from both groups at baseline, two weeks and three months after surgery. Outcome measures for patients include: functional status, nutrition, pain, depression and healthcare consumptions; and for spouses: caregiver satisfaction and difficulties and anxiety.

ELIGIBILITY:
Inclusion Criteria: Patients

* 65 years of age or older
* undergoing a total hip replacement due to arthritis
* live with their spouses
* speak, read and understand Danish without an interpreter
* have their spouses present at the mandatory pre-information meeting in the outpatient facilities.

Inclusion Criteria: Spouses

* presence at the pre-information meeting

Exclusion Criteria: Patients

* They cannot receive home care, be placed in a nursing home or be permanent users of wheelchairs

Exclusion criteria: Both

* Index score at >24 assessed on the Mini-Mental Stats Examination (MMSE)
* Index score of <6 assessed on the Charlson Comorbidity Index

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Functional status/ activities of daily living measured by the Barthel-100, which is a 10-item scale | Three months
Caregiver satisfaction assessed using the 30-item Carer's Assessment of Satisfaction Index (CASI) | Three months

SECONDARY OUTCOMES:
Nutritional improvements measured using the Mini Nutritional Assessment tool (MNA-SF) | Three months
Pain improvements measured using the separate patient-relevant dimension of pain in the Hip Disability and Osteoarthritis Outcome Score (HOOS) | Three months
Depression using the 15-item short form binary reported measurement of the Geriatric Depression Scale (GDS-15) | Three months
Caregiver difficulties assessed through 15 items selected from the 30-item Carer's Assessment of Difficulties (CADI) | Three months
Anxiety assessed using the Generalized anxiety disorder (GAD-7) scale | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Connie B Berthelsen, PhD, Principal Investigator — University of Aarhus